CLINICAL TRIAL: NCT04972149
Title: Cohort Study Comparing Surgeon Stress, Utilization of Surgical Instruments, Surgical Outcomes According to Surgical Approach for Gastrectomy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Other Study IDs: 4-2021-0409
Record Dates: First submitted 2021-07-04; First posted 2021-07-22 (Actual); Last update posted 2021-07-26 (Actual); Status verified 2021-07

CONDITIONS: Gastric Cancer Patients Undergoing Gastrectomy
Keywords: surgeon stress; instrument; outcome; complication

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (6):
- LC: laparoscopic surgery using conventional laparoscopic instruments
- LW: Using wristed laparoscopic instruments (Artisential Maryland dissector, Artisential Fenestrated grasper)
- RC: Conventional robotic surgery
- RSS: Use of single site system for reduced port robotic surgery
- RSP: Use of da Vinci SP system for reduced port robotic surgery
- RRI: A new surgical robot Revo-i developed by Meerae company in Korea

SUMMARY:
A new surgical instrument is supposed to allow surgeon to do surgery with better performance. However, the learning period before getting used to the new instruments is necessary. The surgeon's stress to overcome the learning effect and the surgical outcome was rarely assessed. The comparative analysis of surgical outcome, surgeon's stress, and utilization of instruments for gastrectomy will be performed in prospective cohort study

DETAILED DESCRIPTION:
Before the surgery, all the eligible patients will be explained regarding the study and informed consent will be given. During the surgery, the surgeon will wear heart rate monitoring device to monitor hear rate variability of the surgeon. The surgical procedure will be recorded. After the surgery, morbidity following surgery will be monitored and recorded. At 1 month after surgery, additional morbidity will be recorded.

ELIGIBILITY:
Inclusion Criteria:

Patients with gastric cancer scheduled for gastrectomy

Exclusion Criteria:

Vulnerable subject (illiterate, pregnant)

Max Age: 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with gastric cancer scheduled to undergo gastrectomy in high volume center
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2021-05-18 (Actual); Primary Completion 2022-05-09 (Estimated); Study Completion 2022-07-09 (Estimated)

PRIMARY OUTCOMES:
complication | 1 month after surgery
  One of the most important surgical outcome, complication will be measured at 1 month after surgery

SECONDARY OUTCOMES:
operative time (min) | 1 month after surgery
bleeding(ml) | 1 month after surgery
gas passing(day) | 1 month after surgery
hospital stay(day) | 1 month after surgery
readmission rate(percent) | 1 month after surgery
Heart rate variability of surgeon | during the operation
Duration for each surgical instruments | during the operation
number of use for each surgical instruments | during the operation

CONTACTS AND LOCATIONS:
Overall Officials: Hyoung-Il Kim, Principal Investigator — Yonsei University
Locations (1):
- Severance Hospital, Yonsei University Health System, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Grantcharov PD, Boillat T, Elkabany S, Wac K, Rivas H. Acute mental stress and surgical performance. BJS Open. 2018 Sep 27;3(1):119-125. doi: 10.1002/bjs5.104. eCollection 2019 Feb. PMID 30734023
- [Background] Jeong O, Park YK. Clinicopathological features and surgical treatment of gastric cancer in South Korea: the results of 2009 nationwide survey on surgically treated gastric cancer patients. J Gastric Cancer. 2011 Jun;11(2):69-77. doi: 10.5230/jgc.2011.11.2.69. Epub 2011 Jun 30. PMID 22076206
- [Background] Kim HH, Hyung WJ, Cho GS, Kim MC, Han SU, Kim W, Ryu SW, Lee HJ, Song KY. Morbidity and mortality of laparoscopic gastrectomy versus open gastrectomy for gastric cancer: an interim report--a phase III multicenter, prospective, randomized Trial (KLASS Trial). Ann Surg. 2010 Mar;251(3):417-20. doi: 10.1097/SLA.0b013e3181cc8f6b. PMID 20160637
- [Background] Kim YM, Baek SE, Lim JS, Hyung WJ. Clinical application of image-enhanced minimally invasive robotic surgery for gastric cancer: a prospective observational study. J Gastrointest Surg. 2013 Feb;17(2):304-12. doi: 10.1007/s11605-012-2094-0. Epub 2012 Dec 1. PMID 23207683
- [Background] Kitano S, Iso Y, Moriyama M, Sugimachi K. Laparoscopy-assisted Billroth I gastrectomy. Surg Laparosc Endosc. 1994 Apr;4(2):146-8. PMID 8180768
- [Background] Lee JH, Kim KM, Cheong JH, Noh SH. Current management and future strategies of gastric cancer. Yonsei Med J. 2012 Mar;53(2):248-57. doi: 10.3349/ymj.2012.53.2.248. PMID 22318810
- [Background] Lee S, Kim JK, Kim YN, Jang DS, Kim YM, Son T, Hyung WJ, Kim HI. Safety and feasibility of reduced-port robotic distal gastrectomy for gastric cancer: a phase I/II clinical trial. Surg Endosc. 2017 Oct;31(10):4002-4009. doi: 10.1007/s00464-017-5435-y. Epub 2017 Feb 15. PMID 28205030
- [Background] Liu ZY, Chen QY, Zhong Q, Xie JW, Wang JB, Lin JX, Lu J, Cao LL, Lin M, Tu RH, Huang ZN, Lin JL, Zheng HL, Zheng CH, Huang CM, Li P. Is three-dimensional laparoscopic spleen preserving splenic hilar lymphadenectomy for gastric cancer better than that of two-dimensional? Analysis of a prospective clinical research study. Surg Endosc. 2019 Oct;33(10):3425-3435. doi: 10.1007/s00464-018-06640-7. Epub 2019 Feb 26. PMID 30809728
- [Background] Niitsu H, Hirabayashi N, Yoshimitsu M, Mimura T, Taomoto J, Sugiyama Y, Murakami S, Saeki S, Mukaida H, Takiyama W. Using the Objective Structured Assessment of Technical Skills (OSATS) global rating scale to evaluate the skills of surgical trainees in the operating room. Surg Today. 2013 Mar;43(3):271-5. doi: 10.1007/s00595-012-0313-7. Epub 2012 Sep 1. PMID 22941345
- [Background] Pietrabissa A, Sbrana F, Morelli L, Badessi F, Pugliese L, Vinci A, Klersy C, Spinoglio G. Overcoming the challenges of single-incision cholecystectomy with robotic single-site technology. Arch Surg. 2012 Aug;147(8):709-14. doi: 10.1001/archsurg.2012.508. PMID 22508669
- [Background] Vizza E, Corrado G, Mancini E, Baiocco E, Patrizi L, Fabrizi L, Colantonio L, Cimino M, Sindico S, Forastiere E. Robotic single-site hysterectomy in low risk endometrial cancer: a pilot study. Ann Surg Oncol. 2013 Aug;20(8):2759-64. doi: 10.1245/s10434-013-2922-9. Epub 2013 Mar 7. PMID 23468046
- [Background] Yang SY, Roh KH, Kim YN, Cho M, Lim SH, Son T, Hyung WJ, Kim HI. Surgical Outcomes After Open, Laparoscopic, and Robotic Gastrectomy for Gastric Cancer. Ann Surg Oncol. 2017 Jul;24(7):1770-1777. doi: 10.1245/s10434-017-5851-1. Epub 2017 Mar 29. PMID 28357674
- [Background] Zeng YK, Yang ZL, Peng JS, Lin HS, Cai L. Laparoscopy-assisted versus open distal gastrectomy for early gastric cancer: evidence from randomized and nonrandomized clinical trials. Ann Surg. 2012 Jul;256(1):39-52. doi: 10.1097/SLA.0b013e3182583e2e. PMID 22664559